CLINICAL TRIAL: NCT06546969
Title: A Pilot Study of Chemoimmunotherapy Combined With Hyperthermia and Spatially-Fractionated Radiotherapy in Advanced Biliary Tract Cancer
Brief Title: Chemoimmunotherapy Combined With Hyperthermia and Spatially-Fractionated Radiotherapy in Advanced Biliary Tract Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jason Molitoris, MD PhD, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00109947
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma
Keywords: Chemoimmunotherapy; Spatially Fractionated Radiation Therapy; Deep Hyperthermia
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — Gemcitabine; Cisplatin; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Chemoimmunotherapy + SFRT + Deep Hyperthermia (Experimental): 1. Gemcitabine 1000mg/m2 via intravenous infusion on days 1 and 8 of every 21-day cycle for up to 8 cycles
  2. Cisplatin 25mg/m2 via intravenous infusion on days 1 and 8 of every 21-day cycle for up to 8 cycles
  3. Durvalumab 1500mg via intravenous infusion on day 1 of every 21-day cycle for up to 8 cycles
  4. Deep hyperthermia and spatially-fractionated radiotherapy will be administered to 1 measurable lesion on cycle 2-day 1 and deep hyperthermia alone will be delivered to the same lesion on cycle 3-day 1 and cycle 4-day 1
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Durvalumab; Radiation: Spatially Fractionated RT; Device: Deep Hyperthermia

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2 via intravenous infusion on days 1 and 8 of every 21-day cycle for up to 8 cycles. After the 16 weeks of trial participation, participants will continue chemoimmunotherapy per standard of care.
Drug: Cisplatin — 25mg/m2 via intravenous infusion on days 1 and 8 of every 21-day cycle for up to 8 cycles. After the 16 weeks of trial participation, participants will continue chemoimmunotherapy per standard of care.
Drug: Durvalumab — 1500mg via intravenous infusion on day 1 of every 21-day cycle for up to 8 cycles. After the 16 weeks of trial participation, participants will continue chemoimmunotherapy per standard of care.
Radiation: Spatially Fractionated RT — Administered to 1 measurable lesion on cycle 2-day 1
Device: Deep Hyperthermia — Deep hyperthermia alone will be delivered to the same lesion on cycle 3-day 1 and cycle 4-day 1

SUMMARY:
This study is being done to see if the investigators can improve the outcome of patients with biliary tract cancer that do not qualify for surgery. This study will compare the effects, good and/or bad, of using a combination of standard of care chemoimmunotherapy, with the addition of radiation and deep hyperthermia. In this study, participants will be receiving standard of care chemoimmunotherapy (gemcitabine, cisplatin, and durvalumab), radiation (spatially fractionated radiation therapy), and deep hyperthermia.

Chemoimmunotherapy Chemoimmunotherapy is when chemotherapy drugs are combined with immunotherapy drugs. Chemotherapy uses different drugs to kill or slow the growth of cancer cells, whereas immunotherapy drugs are used to help the immune system attack cancer cells. For this study, the drugs Gemcitabine, Cisplatin, and Durvalumab will be used. Chemoimmunotherapy will be delivered over 4 cycles for this study and can continue longer if the treating physician decides this is appropriate. Each cycle will last 3 weeks.

Spatially fractionated radiation therapy (SFRT) SFRT is a form of radiation therapy that gives a single large dose of radiation to large tumors or tumors that do not qualify for surgery. This is not a standard type of treatment for people with this diagnosis. For this study, participants will be receiving radiation once on day 1 of the second chemoimmunotherapy cycle.

Deep Hyperthermia (HT) Hyperthermia is used in combination with chemoimmunotherapy and radiation treatment in this study. Hyperthermia has the potential to make both chemotherapy and radiation treatments more effective. For this study, participants will receive HT three times: on the first day of cycles 2, 3, and 4 of chemoimmunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
2. Provision of a signed and dated written ICF prior to any mandatory study-specific procedures, sampling, and analyses
3. Age ≥ 21 years at the time of screening
4. Histologically-confirmed, unresectable advanced or metastatic carcinoma of the biliary tract including intrahepatic or extrahepatic cholangiocarcinoma and gallbladder carcinoma
5. No prior systemic therapy for locally advanced, metastatic, or recurrent BTC (prior adjuvant capecitabine therapy is allowed as long as last treatment was ≥ 1 month before enrollment)
6. An ECOG performance status of 0-2 at enrollment
7. At least 1 lesion that qualifies as a RECIST version 1.1 target lesion in the abdomen or pelvis that is amenable to SFRT on contrast enhanced CT or MRI
8. No prior exposure to gemcitabine or platinum-based chemotherapy
9. No prior exposure to anti-PD1 or anti-PDL1 antibodies
10. Adequate organ and marrow function as defined below:

    * Hemoglobin ≥ 9.0 g/dL
    * ANC ≥ 1.5 x 109/L
    * Platelet count ≥ 100 x 109/L
    * Serum bilirubin ≤ 2.5 x upper limit of normal (ULN)
    * Alanine aminotransferase and aspartate aminotransferase ≤ 3 x ULN
    * Measured creatinine clearance > 50 mL/min or calculated creatinine clearance > 50 mL/min as determined by Cockcroft-Gault (using actual body weight)
11. Life expectancy of at least 12 weeks at the time of screening
12. Body weight >30 kg
13. Participants must provide a tumor biopsy taken within 3 years prior to screening
14. Baseline vitals: heart rate of ≤ 90bpm, systolic blood pressure of 140-100mmHg and diastolic of 90-60mmHg

Exclusion Criteria:

1. Ampullary carcinoma
2. History of allogeneic organ transplantation
3. Prior history of radiation to the proposed treatment site
4. Active or prior documented autoimmune or inflammatory disorders with the following exceptions:

   * Participants with vitiligo or alopecia
   * Participants with hypothyroidism stable on hormone replacement
   * Any chronic skin condition that does not requires systemic therapy
   * Participants without an active disease in the last 5 years may be included but only after consultation with the study physician
   * Participants with celiac disease controlled by diet alone
5. Known history or evidence of active, non-infectious pneumonitis
6. Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase the risk of incurring adverse events, or compromise the ability of the participant to give written informed consent
7. Participants with documented myocardial infarction or cerebrovascular accident within 6 months prior to enrollment
8. History of another primary malignancy, except for:

   * Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of investigational product and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease
9. History of leptomeningeal carcinomatosis
10. Active infection including tuberculosis, hepatitis B or hepatitis C. Participants with a past or resolved hepatitis B infection or participants positive for hepatitis C antibody with negative hepatitis C virus RNA on polymerase chain reaction are eligible to enroll. Participants with HIV with undetectable viral load and CD4 cell count ≥200 cells/mm3 are eligible to enroll
11. Any unresolved toxicity per CTCAE version 5.0 grade ≥2 from a previous anticancer therapy, except for alopecia, vitiligo and the laboratory values defined in the inclusion criteria.

    * Participants with grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician
    * Participants with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study physician
12. Untreated brain metastases or spinal cord compression. Participants with suspected brain metastases at screening should have an MRI (preferred) or CT scan, each preferably with IV contrast of the brain prior to study entry
13. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
14. Any concurrent chemotherapy, investigational product, biologic or hormonal therapy for cancer treatment

    • Concurrent use of hormonal therapy for non-cancer related conditions is acceptable
15. Receipt of live attenuated vaccine within 30 days prior to the enrollment
16. Major surgical procedure within 28 days prior to enrollment.
17. Prior locoregional therapy with radioembolization
18. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab with the following exceptions:

    * Intranasal, inhaled, or topical steroids or local steroid injection
    * Systemic corticosteroids at physiologic doses not to exceed 10mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions
19. Participation in another clinical study with an investigational product administered in the last 3 months
20. Concurrent enrollment in another clinical study, unless it is an observational clinical study or during the follow-up period of an interventional study
21. Female participants who are pregnant or breastfeeding or male or female participants of reproductive potential who are not willing to use effective birth control from screening to 180 days after the last dose of gemcitabine/cisplatin or 90 days after the last dose of durvalumab
22. Judgement by the investigator that the participant should not participate in the study if they are unlikely to comply with study procedures, restrictions, and requirements
23. Participants on anti-arrhythmic medication unless they are deemed fit for HT by a consultant cardiologist and there is no increased risk to the patient from HT because of the arrhythmia in the opinion of the treating physician
24. Severe COPD with FEV1 < 50% of expected
25. Participants whose right-to-left pelvic/abdominal dimension is > 49 cm
26. Participants with incorporated metallic implants such as metallic stents, pacemakers or defibrillators, and orthopedic rods and plates of dimensions > 1000/frequency (MHz) aa. Participants who are under any therapy, which by virtue of direct pharmacological action or heat interaction, could influence the intended effects of HT or mask its side effects

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events assessment by CTCAE v5.0 that are grade 3 or higher and related to HT or SFRT | 90 days post final treatment of Deep Hyperthermia
  Determine the safety of combined deep hyperthermia, spatially-fractionated radiotherapy and chemoimmunotherapy in this patient population
  Safety is defined by < 30% rate of grade 3 or higher non-hematologic adverse events possibly or probably related to deep HT or SFRT from cycle 2-day 1 until 90 days post the final deep HT treatment. A rolling safety evaluation will be performed during patient enrollment and termination of the study will occur if any of the below are met
  * Grade 3+ adverse events in more than 1 of the first 3 or 2 of the first 6 patients possibly or probably related to deep HT or SFRT
  * Grade 4+ adverse event in more than 3 total patients possibly or probably related to deep HT or SFRT
  * Grade 5 adverse event in 1 patient where the event is not clearly attributable to the underlying disease or extraneous causes.
Number of participants to receive a minimum of 30 minutes of heating at target temperature (39-43°C) for at least 2 of the planned 3 deep HT treatments | 90 days post final treatment
  Estimate the feasibility of administering combined deep hyperthermia, spatially-fractionated radiotherapy and chemoimmunotherapy for subjects with advanced biliary tract cancer not amenable to surgical resection or definitive local therapy.
  Feasibility is defined as the ability of participants to receive a minimum of 30 minutes of heating at target temperature (39-43°C) for at least 2 of the planned 3 deep HT treatments. A single-group design will be used to obtain a two-sided 95% confidence interval for a single proportion (feasibility). The Exact Clopper-Pearson approach will be used to calculate the confidence interval. The sample proportion is assumed to be 0.7. To produce a confidence interval with a width of no more than 0.5, 15 subjects will be needed.

SECONDARY OUTCOMES:
Radiographic Response Rate | 16 weeks from start of treatment
  Estimate the radiographic response rate at the 16 week imaging timepoint.
  All participants who undergo at least 1 imaging assessment after beginning study will be eligible for radiographic response estimation per RECIST version 1.1 by local radiology review. Baseline CT or MRI scans will be used to select target and non-target lesions.

OTHER OUTCOMES:
Measure absolute number of immune cell subsets | 1 year post completion of accrual
  Exploratory Objective: To assess blood-based correlates of immunity prior to and during treatment for participants on study.
  Immune correlates, through blood sampling, will be measured within 4 weeks of enrollment and approximately every 8 weeks through week 16 to evaluate the degree of immune activation. These analyses will evaluate the absolute number, distribution, and activation status of immune cell subsets
Measure distribution of immune cell subsets | 1 year post completion of accrual
  Exploratory Objective: To assess blood-based correlates of immunity prior to and during treatment for participants on study.
  Immune correlates, through blood sampling, will be measured within 4 weeks of enrollment and approximately every 8 weeks through week 16 to evaluate the degree of immune activation. These analyses will evaluate the absolute number, distribution, and activation status of immune cell subsets
Measure activation status of immune cell subsets | 1 year post completion of accrual
  Exploratory Objective: To assess blood-based correlates of immunity prior to and during treatment for participants on study.
  Immune correlates, through blood sampling, will be measured within 4 weeks of enrollment and approximately every 8 weeks through week 16 to evaluate the degree of immune activation. These analyses will evaluate the absolute number, distribution, and activation status of immune cell subsets

CONTACTS AND LOCATIONS:
Overall Officials: Jason Molitoris, MD, PhD, Principal Investigator — University of Maryland Medical Center / Maryland Proton Treatment Center
Locations (2):
- United States (2):
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No